CLINICAL TRIAL: NCT00967850
Title: Phase III Study of Efficacy and Safety of Intravitreal Bevacizumab in the Treatment of Choroidal Neovascular Membranes Associated to High Myopia
Brief Title: Efficacy and Safety of Intravitreal Bevacizumab in the Treatment of Choroidal Neovascular Membranes Associated to High Myopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOBA-002-2007; EUDRA CT 2007-006785-15
Record Dates: First submitted 2009-08-24; First posted 2009-08-28 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2009-08

CONDITIONS: Myopia; Choroidal Neovascularization
Keywords: High Myopia; Bevacizumab; Photodynamic therapy
MeSH Terms: conditions — Myopia; Choroidal Neovascularization | interventions — Intravitreal Injections; Bevacizumab; Photochemotherapy; Verteporfin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal Bevacizumab (Experimental): Intravitreal injections of bevacizumab
  Interventions: Drug: Intravitreal Injection
- Visudyne (Active Comparator): Photodynamic Therapy with Visudyne
  Interventions: Drug: Photodynamic Therapy (Visudyne)

INTERVENTIONS:
Drug: Intravitreal Injection — Intravitreal injection of 1,25 mg in 0,05 ml
  Other Names: Avastin
  Arms: Intravitreal Bevacizumab
Drug: Photodynamic Therapy (Visudyne) — Photodynamic therapy on day 1 as described in standard clinical guidelines.
  Arms: Visudyne

SUMMARY:
The purpose of this study is to determine the efficacy and safety of intravitreal injections of bevacizumab in High Myopia´s choroidal neovascularization versus the standard treatment of Photodynamic therapy.

DETAILED DESCRIPTION:
Bad response in choroidal neovascularization in High myopia to Photodynamic therapy, which is the current approved treatment for that pathology, and the high incidence of this pathology in these patients, together with the great functional impact in their vision has fostered the search for new therapeutic strategies.

Intravitreal bevacizumab has already been tested in small series of patients with choroidal neovascularization associated to high myopia, whether as first treatment option or after the failure of photodynamic therapy with good results. In the published series an improvement of visual acuity is described after 1-2 injections, with a reduction in the macular edema and a good safety profile.

The lack of published trials that describe the efficacy of frequency of treatment in this pathology is the main reason for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* High Myopia with one of the following:

  * 6 or more sphere diopters in the study eye
  * Axial length of the eye greater than 26 millimeters
* Active subfoveal/juxtafoveal choroidal neovascularization confirmed by Fluorescein angiography and Ocular coherence tomography.
* Visual acuity loss of less than 6 months of evolution related to the neovascular lesion, as stated by investigator´s opinion.
* Patients previously treated with Photodynamic therapy are allowed to participate as long as the last treatment has been performed more than 3 months upon entering the study.
* Signed informed consent.
* Signed data protection consent.
* Women of childbearing potential must provide a negative pregnancy test at inclusion and must commit to the use of a contraceptive treatment during the whole study.

Exclusion Criteria:

* Previous vitrectomy surgery in the study eye.
* Tractional maculopathy and/or epiretinal membrane evaluated by Ocular coherence tomography.
* Opacities that may not allow correct fundus assessment.
* Lack of integrity of the posterior lens capsule in pseudoaphakic patients.
* Patients that may not want/be able to complete the study, based in the investigator opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Improvement in Visual Acuity assessed by ETDRS | Every month during first year - Every three months during the second year

SECONDARY OUTCOMES:
Central macular thickness with Ocular Coherence Tomography | Every month during first year - Every three months during the second year
Complications that may arise from intravitreal injection | Every treatment visit - Once per month during the first 3 months. Reteatments depending on Visual acuitiy evolution and retinal thickness

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Pastor Jimeno, MD, PhD, Principal Investigator — IOBA - Instituto Universitario de Oftalmobiología Aplicada
Locations (7):
- Spain (7):
  - INGO, Santiago de Compostela, La Coruña
  - Hospital General Reina Sofía, Espinardo, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmológico de Alicante, Alicante
  - Hospital de la Vall d´Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - IOBA - Instituto Universitario de Oftalmobiología Aplicada, Valladolid